CLINICAL TRIAL: NCT06106386
Title: The Impact of Using Cold Irrigation on Postoperative Endodontic Pain and Substance P Level: a Randomized Clinical Trial
Brief Title: The Effect of Different Intraradicular Cryotherapy on Post-operative Pain and the Level of Substance P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maram Obeid, Professor of Endodontics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20720
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Pain; Inflammation
Keywords: Cryotherapy; Substance P; Apical periodontitis; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative; Inflammation; Periapical Periodontitis | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Conventional root canal treatment is done and irrigation will be done with 2.5% room temperature sodium hypochlorite
- Cryotherapy Group (Experimental): Root canal treatment is done and irrigation is done with cooled sodium hypochlorite ( 2- 4°C) through out the visits and final flush with 2- 4°C cold saline will be used for 5 minutes.
  Interventions: Other: cryotherapy
- Final Flush group (Active Comparator): Root canal treatment is done and irrigation is done with sodium hypochlorite at room temperature through out the visits then final flush with 2- 4°C cold saline will be used for 5 minutes.
  Interventions: Other: cryotherapy

INTERVENTIONS:
Other: cryotherapy — Cooling of irrigation
  Arms: Cryotherapy Group; Final Flush group

SUMMARY:
The aim of this clinical trial is to evaluate the effect of using intra-radicular cryotherapy technique in the form of irrigation with cold sodium hypochlorite

The main questions to answer are:

1. Does Postoperative pain is different between the three groups?
2. Does level of substance P different between the three groups ?

DETAILED DESCRIPTION:
* The patients will be randomly divided into three groups Group 1: control group (n=25) Regular root canal treatment with regular irrigant will be used. Group 2: (n=25) Intraradicular cryotherapy will be performed where :
* Normal root canal treatment will be done with irrigation using sodium hypochlorite cooled to 2°C continuously during our mechanical instrumentation. Then a final flush will be done with cold saline 2°C for 5 minutes. Group 3: (n=25) Normal root canal treatment will be done with irrigation using sodium hypochlorite at room temperature during our mechanical instrumentation. Then a final flush will be done with cold saline 2°C for 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will be diagnosed with symptomatic apical periodontitis
* Single-rooted premolars (radiographically and clinically assessed)
* Medically free patients.
* Teeth with mature apex

Exclusion Criteria:

* Patients with other pulpal diagnosis.
* Medically compromised patients.
* Pregnant females.
* Patients taking analgesics or anti-inflammatory drugs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Level of post operative pain | after 6 hours, 24 hours, 48 hours, 72 hours
  On visual analogue scale (VAS) questionnaire, patients will report their level of pain 0° refers for no pain, and the 100° degree refers for unbearable pain

SECONDARY OUTCOMES:
Level of substance P | After access cavity, after finishing mechanical perpetration, before obturation(after 3 days)
  apical fluid sample will be taken using sterilized, medium sized paper point (Diadent Korea, Seoul, Korea) will be inserted into the periapical area and left in place for 30 seconds and the sample will be placed into a 1.5-mL Eppendorf tube containing 100 _L of Tris-HCl buffer, pH 7.5, with 0.15 M NaCl and 1 mM CaCl2; the tubes will be placed on a shaker at room temperature for 3 hours and then stored at -70°C

CONTACTS AND LOCATIONS:
Overall Officials: Maram F Obeid, Professor, Study Director — Faculty of dentistry Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: 2025

REFERENCES:
- [Derived] Sharaf RMA, Abdelrahman TY, Obeid MF. The impact of using cold irrigation on postoperative endodontic pain and substance P level: a randomized clinical trial. Odontology. 2025 Jun 18. doi: 10.1007/s10266-025-01131-3. Online ahead of print. PMID 40533695